CLINICAL TRIAL: NCT01709877
Title: Randomised Non-inferiority Trial of Laparoscopic Cholecystectomy Performed With EndoCone Single Port Versus Conventional Multi-port Laparoscopic Approach Using Clinical, PROMS and Health Economic Endpoints
Brief Title: EndoCone Single Port Versus Conventional Multi-port Laparoscopic Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Collaborators: Regione Toscana (Unknown); Scuola Superiore Sant'Anna di Pisa (Other); Università di Pisa (Unknown)
Responsible Party: Principal Investigator, Franco Mosca, Prof., Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOUP_1; RF-2009-1535329 (Other: Ministero della Salute - Direzione Generale della Ricerca Scientifica e Tecnologica; Regione Toscana)
Record Dates: First submitted 2012-10-17; First posted 2012-10-18 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Gallstones
Keywords: Multiport laparoscopy; Single Port Laparoscopy; Symptomatic Gallstones
MeSH Terms: conditions — Gallstones | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional multiport laparoscopic cholecystectomy (Active Comparator): Standard laparoscopic cholecystectomy performed by the traditional multiport technique
  Interventions: Procedure: Cholecystectomy
- Single port laparoscopic cholecystectomy (Experimental): Laparoscopic cholecystectomy performed using the reusable ENDOCONE system with dedicated curved coaxial instruments
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Multiport and single-port laparoscopic cholecystectomy in patient with symptomatic gallstone disease

SUMMARY:
Its main objective is to evaluate the clinical outcome (including patient reported outcomes) and health economic assessment (HTA) of a new re-usable system for Single Port Laparoscopic Surgery - ENDOCONE SYSTEM developed by Prof Cuschieri by undertaking a randomised controlled prospective clinical trial (RCT) on specific operations performed (on a random allocation basis) by either the traditional multi-port laparoscopic approach or the Single Port- ENDOCONE system by Karl Storz. To this effect, 300 patients meeting the trial inclusion criteria will be randomised over a three year period to have the operation by either of the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic gallstone disease
* ASA I/II
* Age between 18 and 80 years

Exclusion Criteria:

* ASA III or more
* significant co-morbid cardiovascular, neurological diseases, diabetics and chronic obstructive airway disease
* patients with previous history of invasive cancer
* patients with previous surgery
* patients requiring urgent/emergency interventions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-07 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | During the intervention
  1 = if the intervention is converted to open surgery 0 = if the intervention is completed using standard laparoscopy or single port
Morbidity | 30 days
  1 = if the patient has surgical complications 0 = no complications
Mortality | 30 days

SECONDARY OUTCOMES:
Postoperative course | 1 week
  pain, measured using 1) visual linear analogue scale and 2) analgesic administration
Duration of hospital stay | 6 days
  Date of the operation Date of hospital discharge
Return of bowel function | 12, 24, 48 hours
  Passage of flatus and/or bowel motion

CONTACTS AND LOCATIONS:
Overall Officials: Franco Mosca, Prof, MD, Principal Investigator — AOUP; Alfred Cuschieri, Prof, MD, Principal Investigator — Scuola Superiore Sant'Anna di Pisa
Locations (4):
- Italy (4):
  - Ospedale San Donato, Arezzo, AR
  - Ospedale Campo di Marte, Lucca, LU
  - Ospedinale di Cisanello, Pisa, PI
  - Ospedale Felice Lotti, Pontedera, PI